CLINICAL TRIAL: NCT01956760
Title: A Randomized Controlled Clinical Trial to Evaluate Effectiveness of Acupuncture on Insomnia
Brief Title: Effects of Acupuncture and Intradermal Acupuncture on Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Kyunghee University (Other)
Responsible Party: Principal Investigator, Sun Yong Chung, assistant professor, Kyunghee University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KHNMC-OH-IRB 2011-015
Record Dates: First submitted 2013-09-05; First posted 2013-10-08 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Insomnia
Keywords: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental): Acupuncture and intradermal acupuncture The acupuncture was applied at 5 acupoints(HT7 Shenmen, PC6 Neiguan, SP6 Sanyinjiao, KI6 Zhaohai, BL62 Shenmai) 3 times in a week. It was performed by a certified practitioner with sterile needles (0.25*40.0mm). The needles were inserted at least 10.0mm deep through the skin and maintained for 20 minutes The intradermal acupuncture was applied at the same acupoints, immediately after the acupuncture needles were removed. It was performed by the same practitioner with sterile needles (0.20*8.0mm).attached to skin tape (10.0*10.0mm). The needles were inserted 3.0~5.0mm deep and maintained for 48~72 hours
  Interventions: Other: Acupuncture and intradermal acupuncture
- Placebo Acupuncture (Placebo Comparator): Placebo acupuncture and placebo intradermal acupuncture The acupuncture was applied 3 times in a week at 2 sham points on the wrist and 3 sham points on the ankle, approximately 1cm lateral to the acupoints. It was performed by a certified practitioner with sterile needles (0.25*40.0mm). The needles were inserted at least 10.0mm deep through the skin and maintained for 20 minutes The intradermal acupuncture was applied at the same sham points, immediately after the acupuncture needles were removed. It was performed by the same practitioner with sterile needles (0.20*8.0mm).attached to skin tape (10.0*10.0mm). The needles were inserted 3.0~5.0mm deep and maintained for 48~72 hours

INTERVENTIONS:
Other: Acupuncture and intradermal acupuncture — The acupuncture was applied at 5 acupoints(HT7 Shenmen, PC6 Neiguan, SP6 Sanyinjiao, KI6 Zhaohai, BL62 Shenmai) 3 times in a week. It was performed by a certified practitioner with sterile needles (0.25*40.0mm). The needles were inserted at least 10.0mm deep through the skin and maintained for 20 minutes The intradermal acupuncture was applied at the same acupoints, immediately after the acupuncture needles were removed. It was performed by the same practitioner with sterile needles (0.20*8.0mm).attached to skin tape (10.0*10.0mm). The needles were inserted 3.0~5.0mm deep and maintained for 48~72 hours
  Arms: Acupuncture

SUMMARY:
The aim of this clinical study is to observe the therapeutic effect of acupuncture and intradermal acupuncture in the treatment of insomnia

Participants were randomized into the acupuncture group and control group. Both groups were treated 3 times in a week and assessed before and after the treatment.

Hypothesis :

1. Acupuncture group will produce superior effect in the treatment of insomnia compared with control group.
2. Acupuncture group will produce superior improvement in anxiety, depression, quality of life, sleep log, recognition, attention, and memory.

DETAILED DESCRIPTION:
The acupuncture group is received acupuncture and intradermal acupuncture therapy at 5 acupoints on wrist and ankle. The control group is received same treatment at 5 sham points approximately 1cm lateral to the acupoints.

Except for the location of acupuncture points, all details of treatment are same between acupuncture group and control group. A certified practitioner treat both groups 3 times in a week. The acupuncture inserted into the skin for 20 minutes and the intradermal acupuncture inserted and fixed on the same points for 48~72 hours.

Severity of insomnia, anxiety, depression, quality of life, recognition, attention, and memory are assessed at the baseline, after the last treatment and at a week after the end of last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the age of 18years and 65 years.
* Diagnosed as having Insomnia using Pittsburgh Sleep Quality Index(PSQI score>5).
* Have no problems with communication (for example, reading, writing, listening, speaking).
* Provided written informed consent.

Exclusion Criteria:

* Regular medication, Herbal medication or health functional food for treating insomnia
* Presence of major neuropsychiatric disorder (for example, mental retardation, psychosis and severe mood disorder)
* Presence of inflammatory skin disease on the acupuncture site
* Presence of bleeding disorders or takes anticoagulant
* Presence of severe physical diseases that may preclude the safe use of acupuncture
* Enrolled in another clinical study in the past 1 month
* Pregnancy or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in ISI(Insomnia Severity Index) at 1 week | baseline and 1 week

SECONDARY OUTCOMES:
Change from Baseline in ISI(Insomnia Severity Index) at 2 weeks | baseline and 2 weeks
  Follow-up
Change from Baseline in STAI(State-Trait Anxiety Inventory) at 1 week | baseline and 1 week
Change from Baseline in STAI(State-Trait Anxiety Inventory) at 2 weeks | baseline and 2 weeks
  Follow-up
Change from Baseline in BDI(Beck Depression Inventory) at 1 week | baseline and 1 week
Change from Baseline in BDI(Beck Depression Inventory) at 2 weeks | baseline and 2 weeks
  Follow-up
Change from Baseline in PSQI(Pittsburgh Sleep Quality Index) at 1 week | baseline and 1 week
Change from Baseline in PSQI(Pittsburgh Sleep Quality Index) at 2 weeks | baseline and 2 weeks
  Follow-up
Change from Baseline in Sleep Logs at 1 week | baseline and 1 week
  Sleep onset latency, Total sleep time, Wake time after sleep onset and Sleep efficiency
Change from Baseline in Sleep Logs at 2 week | baseline and 2 weeks
  Sleep onset latency, Total sleep time, Wake time after sleep onset and Sleep efficiency
  Follow-up
Change from Baseline in WHOQOL-Bref at 2 weeks | baseline and 2 weeks
Change from Auditory Verbal Learning Test at 1 week | baseline and 1 week
Change from Baseline in Auditory Verbal Learning Test at 2 weeks | baseline and 2 weeks
  Follow-up
Change from Digit Span Test at 1 week | baseline and 1 week
Change from Digit Span Test at 2 weeks | baseline and 2 weeks
  Follow-up
Change from Spectral analysis EEG at 1 week | baseline and 1 week
Change from Spectral analysis EEG at 2 weeks | baseline and 2 weeks
  Follow-up
Change from Auditory ERP at 1 week | baseline and 1 week
Change from Auditory ERP at 2 weeks | baseline and 2 weeks
  Follow-up
Change from Heart Rate Variability at 1 week | baseline and 1 week
Change from Heart Rate Variability at 2 weeks | baseline and 2 weeks
  Follow-up

CONTACTS AND LOCATIONS:
Overall Officials: SUNYONG CHUNG, ph.D, Principal Investigator — Kyunghee University
Locations (1):
- HYUNG-HEE UNIVERSITY HOSPITAL at GANGDONG, Seoul, South Korea

REFERENCES:
- [Derived] Han KH, Kim SY, Chung SY. Effect of acupuncture on patients with insomnia: study protocol for a randomized controlled trial. Trials. 2014 Oct 23;15:403. doi: 10.1186/1745-6215-15-403. PMID 25342100